CLINICAL TRIAL: NCT02231281
Title: A Randomized, Open-label Trial to Compare the Efficacy and Safety of Early Initiation of cART With or Without Autologous HIV-1 Specific Cytotoxic T Lymphocyte (CTL) Infusion in Treatment-Naïve Acute HIV-1 Infected Adults
Brief Title: Early cART and cART in Combination With Autologous HIV-1 Specific Cytotoxic T Lymphocyte (CTL) Infusion in The Treatment of Acute HIV-1 Infected Adults
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Yongtao Sun, MD, PhD (Other)
Collaborators: Tang-Du Hospital (Other); National Center for AIDS/STD Control and Prevention, China CDC (Other Government); Beijing YouAn Hospital (Other); China Medical University, China (Other); Shandong Province Centers for Disease Control and Prevention (Other); Zhejiang University (Other); First Affiliated Hospital of Guangxi Medical University (Other)
Responsible Party: Sponsor-Investigator, Yongtao Sun, MD, PhD, Director of Department of Infectious Diseases, Tang-Du Hospital
Organization: Tang-Du Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014ZX10001002-001; 2014ZX10001002-001 (Other Grant/Funding Number: National Science and Technology Major Project of China during the "12th Five-Year Plan")
Record Dates: First submitted 2014-08-26; First posted 2014-09-04 (Estimated); Last update posted 2018-04-26 (Actual); Status verified 2018-04

CONDITIONS: Acute HIV Infection
Keywords: HIV Infections; Acquired Immunodeficiency Syndrome; Immunologic Deficiency Syndromes; Immune System Diseases; Lentivirus Infections; Retroviridae Infections; Virus Diseases; RNA Virus Infections; Sexually Transmitted Diseases, Viral; Slow Virus Diseases; Therapeutic Uses; Pharmacologic Actions; Antiretroviral therapy; Early therapy
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; Immunologic Deficiency Syndromes; Immune System Diseases; Lentivirus Infections; Retroviridae Infections; Virus Diseases; RNA Virus Infections; Sexually Transmitted Diseases, Viral; Slow Virus Diseases | interventions — Tenofovir; Zidovudine; Lamivudine; Lopinavir; Ritonavir; lopinavir-ritonavir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- cART(TDF/AZT+3TC+LPV/r) (Experimental): cART(TDF/AZT+3TC+LPV/r)
  Interventions: Drug: cART(TDF/AZT+3TC+LPV/r)
- CTL infusion (Experimental): cART plus autologous HIV-1 specific cytotoxic T lymphocyte (CTL) infusion
  Interventions: Drug: cART(TDF/AZT+3TC+LPV/r); Procedure: CTL infusion

INTERVENTIONS:
Drug: cART(TDF/AZT+3TC+LPV/r) — Standard antiretroviral therapy for HIV infection
  Other Names: Tenofovir Disoproxil Fumarate; Zidovudine; Lamivudine; Lopinavir/ritonavir (Kaletra)
Procedure: CTL infusion — cART(TDF/AZT+3TC+LPV/r) plus autologous HIV-1 specific cytotoxic T lymphocyte (CTL) infusion
  Arms: CTL infusion

SUMMARY:
The purpose of this study is to assess the ability of the early initiation of cART or cART in combination with autologous HIV-1 specific cytotoxic T lymphocyte (CTL) infusion to achieve a post-treatment control among treatment-naïve acute HIV-infected adults.

DETAILED DESCRIPTION:
Although combined antiretroviral therapy (cART) can suppress HIV-1 replication to a very low level in the blood, but it cannot eliminate latent viral reservoirs, and need lifelong adherence to expensive regimens that have potential side effects. Increasing evidence indicates that early antiretroviral therapy for recently HIV-infected patients results in slower progression of HIV disease and represent a unique opportunity to interfere with either the quantities or qualities of persistent reservoirs of replication-competent virus. However, the time course before the interruption of cART is unclear. This study will compare the virological and immunological outcomes and HIV latency of recently infected adults who receive cART or cART in combination with autologous HIV-1 CTL infusion for different periods.

The study will last 120 weeks. Participants will be randomly assigned to either the cART or the cART plus autologous HIV-1 CTL infusion arm of one of three cohorts. The three cohorts will differ in the period of cART given. Cohort 1, Cohort 2 or Cohort 3 will receive cART (Zidovudine (AZT)/Tenofovir disoproxil fumarate (TDF) +Lamivudine (3TC） + Lopinavir / Ritonavir （LPV/r)） for 48, 72 or 96 weeks, respectively. After 48, 72 or 96 weeks, cART will be interrupted respectively. Study visits will occur at study entry, Week 4 and 12, and every 12 weeks thereafter through treatment interruption, then every 4 weeks through 12 weeks later, then every 12 weeks through Week 120. At each study visit, a physical exam, blood collection, and completion of an adherence questionnaire will occur. Clinical, virological, and immunological evaluations and HIV latency examination will be performed at most study visit.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of acute HIV infection (meets one of following criteria)

   1. Negative for anti-HIV test formerly, but with an anti-HIV serological conversion within 6 months
   2. Detection of plasma HIV RNA by RT-PCR in the absence of HIV antibody
   3. Low-level of anti-HIV for BED HIV-1 capture enzyme immuno assay (BED-CEIA), optical density (OD)<0.6, only for B subtype)
   4. Uncertain for an anti-HIV test, with an increasing anti-HIV level for repeated test within two weeks
   5. A patient with a report of recent risk behavior in association with symptoms and signs of the acute retroviral syndrome, as well as a positive for HIV antigen detection and less than 4 bands in a Western blot assay
2. Ability, willingness to give informed consent
3. Able, willing to adhere to therapy and adherent to ART
4. Able, willing to comply with time requirements for study visits and evaluations

Exclusion Criteria:

1. Chronic HIV - 1 infection
2. Any evidence of an active AIDS-defining opportunistic infection
3. Screening detects the following results:HGB<90g/L、WBC< 2 x 10E9/L、PLT< 75 x 10E9/L、hemodiastase>2 x ULN、Scr>1.5 x ULN、ALT/AST/ALP> 3 xULN、TbiL>2 xULN、CK>2 xULN、CCr<60ml/min
4. A personal history of clinically significant cardiac disease, symptomatic or asymptomatic arrhythmias, syncopal episodes, or additional risk factors for torsades de points
5. History of chronic kidney disease
6. History of malignancy or transplantation, including skin cancers or Kaposi sarcoma
7. History of Severe peptic ulcer
8. History of alcoholism and drug abuse
9. Receipt of immunomodulating agents, immunization or systemic chemotherapeutic agents within 28 days prior to screening
10. Women who are pregnant or breastfeeding, or with a positive pregnancy test during screening or Women of Child Bearing Potential (WOCBP) who are unwilling or unable to use an acceptable method of contraception to avoid pregnancy for the entire study period
11. Have contraindications to cART
12. Other condition that does not fit to participate in this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2014-08 (Actual); Primary Completion 2018-08 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in HIV DNA quantification at the interruption of cART | 48 weeks for Cohort 1, 72 weeks for Cohort 2, 96 weeks for Cohort 3
  HIV DNA detection includes total HIV DNA, integrated HIV DNA , 2-long terminal repeat （LTR） HIV DNA in resting CD4+T cell subsets.
Number of patients who achieve virological remission | 72 weeks for Cohort 1, 96 weeks for Cohort 2, 120 weeks for Cohort 3
  Virological remission is defined as undetectable of plasma HIV RNA for 24 weeks after the interruption of cART.

SECONDARY OUTCOMES:
Number of patients who occur any grade 3 or 4 (clinical or laboratory) adverse events | 120 weeks
Number of patients who need to initiate late treatment | 120 weeks
  Late treatment is defined cART should be administered according to local HIV treatment guidelines.
Time from cART interruption to virological relapse (plasma viral load more than 50 copies/mL) | 120 weeks
HIV-1 specific CD4+ and CD8+ T cell responses at week 120 | 120 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yongtao Sun, M.D., Ph.D., Principal Investigator — Department of Infectious Diseases, Tangdu Hospital, The Fourth Military Medical University
Locations (7):
- China (7):
  - Beijing You'an Hospital, Capital Medical University, Beijing, Beijing Municipality
  - National Center for STD and AIDS Control and Prevention, Chinese Center for Disease Control and Prevention, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - China Medical University, Shenyang, Liaoning
  - Department of Infectious Diseases, Tangdu Hospital, The Fourth Military Medical Universit, Xi'an, Shaanxi
  - Shandong Center for Disease Control and Prevention, Jinan, Shandong
  - Zhejiang University, Hangzhou, Zhejiang